CLINICAL TRIAL: NCT01423123
Title: A Phase I Dose-Escalation Study Evaluating the Combination of Weekly Paclitaxel With Neratinib and Trastuzumab in Women With Metastatic HER2-positive Breast Cancer
Brief Title: Combination of Weekly Paclitaxel With Neratinib and Trastuzumab in Women With Metastatic HER2-positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FB-8; WS1554503 (Other: Pfizer Inc.)
Record Dates: First submitted 2011-08-19; First posted 2011-08-25 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
Keywords: Paclitaxel; Trastuzumab; Neratinib; Breast Cancer; HER2-positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab; neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neratinib (Experimental): Paclitaxel (80 mg/m2 IV on days 1, 8, and 15 every 28 days) and trastuzumab (4 mg/kg/ loading dose, then 2 mg/kg) IV weekly beginning on day 1 of paclitaxel, neratinib orally daily beginning on day 1 of paclitaxel until disease progression.
  Interventions: Drug: Paclitaxel; Biological: trastuzumab; Drug: Neratinib

INTERVENTIONS:
Drug: Paclitaxel — 80 mg/m2 IV on days 1, 8, and 15 every 28 days until disease progression.
Biological: trastuzumab — 4 mg/kg IV loading dose, then 2 mg/kg IV weekly until disease progression.
Drug: Neratinib — Dose level 1: 120 mg/day orally; Dose level 2: 160 mg/day orally; Dose level 3: 240 mg/day orally; Dose level 4: 200 mg/day orally.

SUMMARY:
The FB-8 study is designed as an open label, single arm, Phase I dose-escalation study evaluating the combination of weekly paclitaxel with neratinib and trastuzumab in women with metastatic, HER2-positive breast cancer. The primary aim of this study is to determine the safety and tolerability of the three-drug combination.

DETAILED DESCRIPTION:
Patients will receive concurrent therapy with paclitaxel (80 mg/m2 IV on days 1, 8, and 15 of a 28-day cycle), trastuzumab (4 mg/kg IV loading dose, then 2 mg/kg IV weekly), and neratinib. The neratinib dose-escalation will include 4 dose levels (120 mg, 160 mg, 200 mg, and 240 mg) as a daily oral dose.

The neratinib dose-escalation for the study will proceed on the basis of dose-limiting toxicity (DLT) during cycle 1. DLT will be defined as the occurrence of 1 or more of the following events during cycle 1: any grade diarrhea that is associated with fever or dehydration; grade 3 diarrhea lasting more than 2 days on optimal medical therapy; grade 4 diarrhea of any duration; grade 3 or 4 neutropenia associated with fever; grade 4 neutropenia lasting more than 7 days; grade 4 thrombocytopenia; grade 3 or 4 non-hematological toxicity; or any toxicity-related delay of more than 2 weeks to initiate cycle 2. Patients will be enrolled at the next dose level when all evaluable patients at the same dose level have completed the first treatment cycle. Enrolled patients will remain on the assigned dose level treatment until toxicity or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Co-morbid conditions should be taken into consideration, but not the diagnosis of metastatic breast cancer.
* Patients of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy and for at least 6 months after the last dose of study therapy.
* The ECOG performance status must be 0, 1, or 2.
* Patients must have the ability to swallow oral medication.
* Patients must have histologic or cytologic confirmation of the diagnosis of invasive adenocarcinoma of the breast.
* There must be documentation that the patient has evidence (measurable or non-measurable) of metastatic breast cancer. Histologic confirmation of metastatic disease is not required.
* Patients must have ER analysis performed on the primary tumor prior to study entry. If ER analysis is negative, then PgR analysis must also be performed. (Patients are eligible with either hormone receptor-positive or hormone receptor-negative tumors.)
* Breast cancer must be determined to be HER2-positive prior to study entry. Assays using FISH or CISH require gene amplification. Assays using IHC require a strongly positive (3+) staining score.
* At the time of study entry, blood counts performed within 4 weeks prior to study entry must meet the following criteria: ANC must be greater than or equal to 1000/mm3; Platelet count must be greater than or equal to 100,000/mm3; Hemoglobin must be greater than or equal to 9 g/dL
* The following criteria for evidence of adequate hepatic function performed within 4 weeks prior to study entry must be met: total bilirubin must be less than or equal to 1.5 x ULN; AST and ALT must be less than or equal to 2.5 x ULN for the lab or less than or equal to 5 x ULN if liver metastasis
* Serum creatinine performed within 4 weeks prior to study entry must be less than or equal to 1.5 x ULN for the lab.
* The LVEF assessment by 2-D echocardiogram or MUGA scan performed within 90 days prior to study entry must be greater than or equal to 50% regardless of the facility's LLN.

Exclusion Criteria:

* Previous therapy with neratinib for any malignancy.
* Symptomatic brain metastases or brain metastases requiring chronic steroids to control symptoms.
* Active hepatitis B or hepatitis C with abnormal liver function tests.
* Intrinsic lung disease resulting in dyspnea.
* Active infection or chronic infection requiring chronic suppressive antibiotics.
* Malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease or condition significantly affecting gastrointestinal function.
* Persistent greater than or equal to grade 2 diarrhea regardless of etiology.
* Sensory or motor neuropathy greater than or equal to grade 2, as defined by the NCI CTCAE v3.0.
* Conditions that would prohibit intermittent administration of corticosteroids for paclitaxel premedication.
* Chronic daily treatment with corticosteroids with a dose of greater than or equal to 10 mg/day methylprednisolone equivalent (excluding inhaled steroids).
* Uncontrolled hypertension defined as a systolic BP greater than 150 mmHg or diastolic BP greater than 90 mmHg, with or without anti-hypertensive medications (Patients with hypertension that is well controlled on medication are eligible.)
* Cardiac disease (history of and/or active disease) that would preclude the use of any of the drugs included in the treatment regimen. This includes but is not confined to: Active cardiac disease: symptomatic angina pectoris within the past 90 days that required the initiation of or increase in anti-anginal medication or other intervention; ventricular arrhythmias except for benign premature ventricular contractions; supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; conduction abnormality requiring a pacemaker; valvular disease with documented compromise in cardiac function; and symptomatic pericarditis. History of cardiac disease: myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LV function; history of documented CHF; and documented cardiomyopathy
* Other nonmalignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow up.
* Pregnancy or lactation at the time of study entry. (Note: Pregnancy testing should be performed within 14 days prior to study entry according to institutional standards for women of childbearing potential.)
* The investigator should assess the patient to determine if she has any psychiatric or addictive disorder or other condition that, in the opinion of the investigator, would preclude her from meeting the study requirements.
* Use of any investigational agent within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the three-drug combination | Through 6 months after last dose
  Number of patients experiencing dose limiting toxicities (DLT).

SECONDARY OUTCOMES:
Overall response rate | Measured at 24 weeks from start of therapy.
  Number of patients with disappearance of all target lesions; Number of patients with at least a 30% decrease in the sum of the longest diameter (LD) of target lesions; patients with neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as a reference the smallest sum LD since baseline.
Progression-free interval | Time to disease progression up to 15 months.
  Number of patients with at least a 20% increase in the sum of the LD of target lesions, taking as a reference the smallest sum LD recorded since baseline or the appearance of one or more new lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (4):
- United States (4):
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NSABP Foundation, Inc., Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - West Virginia University Hospitals, Morgantown, West Virginia

REFERENCES:
- [Result] Jankowitz RC, Abraham J, Tan AR, Limentani SA, Tierno MB, Adamson LM, Buyse M, Wolmark N, Jacobs SA. Safety and efficacy of neratinib in combination with weekly paclitaxel and trastuzumab in women with metastatic HER2-positive breast cancer: an NSABP Foundation Research Program phase I study. Cancer Chemother Pharmacol. 2013 Dec;72(6):1205-12. doi: 10.1007/s00280-013-2262-2. PMID 24077916